CLINICAL TRIAL: NCT01683578
Title: Effects of Variable Tidal Volumes During Open Abdominal Surgery on Lung Function and Systemic Inflammation
Brief Title: Protective Variable Ventilation for Open Abdominal Surgery
Acronym: PROVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PulmEngineering-2012-01
Record Dates: First submitted 2012-09-03; First posted 2012-09-12 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Development of Pulmonary Dysfunction Following Open Abdominal Surgery
Keywords: mechanical ventilation; lung function; abdominal surgery, open; systemic inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Variable Ventilation (Active Comparator): Variable tidal volumes with mean at 8 mL/kg of predicted body weight
  Interventions: Other: Variable Ventilation
- Non-variable Ventilation (No Intervention): Conventional mechanical ventilation with tidal volume 8 mL/kg of predicted body weight

INTERVENTIONS:
Other: Variable Ventilation
  Arms: Variable Ventilation

SUMMARY:
Variable ventilation has been shown to improve lung function and reduce lung damage as well as inflammation in different models of the acute respiratory distress syndrome. Also, variable ventilation is able to recruit lungs. The present study will investigate whether variable as compared to non-variable ventilation improves post-operative lung function and reduces systemic inflammation in patients submitted to open abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective open abdominal surgery
* ASA classification 2-3
* age between 18 und 85 yrs
* expected duration of surgery > 3 h
* expected extubation in the operation room
* written informed consent

Exclusion Criteria:

* chronic lung disease (except to COPD stadium I and II, and asthma)
* Body Mass Index (BMI) > 40
* allergy to one of the drugs to be used for general anesthesia
* participation in another interventional trial within 4 weeks before enrollment
* addiction or any other disease that may interfere with the capacity of giving informed consent
* pregnant or breastfeeding women
* women in reproductive age, except to those who fulfill one of the following:

  * post-menopause (12 months natural amenorrhoea, or 6 months amenorrhoea and serum FSH > 40 mlU/ml
  * post-operative (6 weeks after two-sided ovariectomy)
  * routine and correct use of anticonceptional methods with failure rate < 1 % per year
  * sexually not active
  * vasectomy of the partner
* indication of low compliance with the protocol
* contraindication for MRI examination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | Preoperative until 5th postoperative day
  Forced vital capacity is assessed on the first postoperative day

SECONDARY OUTCOMES:
Arterial partial CO2 pressure | Preoperative until 5th postoperative day
  PacO2 on the first postoperative day
Peak expiratory flow | Preoperative until 5th postoperative day
Forced expiratory volume after 1 sec | Preoperative until 5th postoperative day
  Forced expiratory volume after 1 sec (FEV1) on first postoperative day
PaO2/FIO2 | Preoperative until 5th postoperative day
  PaO2/FIO2 during the intraoperative period
Distribution of ventilation | Preoperative until 5th postoperative day
  Distribution of ventilation in lungs
Atelectasis | Preoperative until 5th postoperative day
  Amount of lung atelectasis on the first postoperative day
Postoperative pulmonary complications | Preoperative until discharge from hospital
  Development of postoperative pulmonary complications
Inflammation markers | Preoperative until 5th postoperative day
  Concentrations of interleukine(IL)-6, IL-8 and tumor necrosis factor(TNF)-alpha in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Gama de Abreu, MD, PhD, Principal Investigator — Klinikum Ludwigshafen
Locations (1):
- Department of Anesthesiology and Intensive Care, University Hospital Carl Gustav Carus, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Spieth PM, Guldner A, Uhlig C, Bluth T, Kiss T, Conrad C, Bischlager K, Braune A, Huhle R, Insorsi A, Tarantino F, Ball L, Schultz MJ, Abolmaali N, Koch T, Pelosi P, Gama de Abreu M; PROtective Ventilation (PROVE) Network. Variable versus conventional lung protective mechanical ventilation during open abdominal surgery (PROVAR): a randomised controlled trial. Br J Anaesth. 2018 Mar;120(3):581-591. doi: 10.1016/j.bja.2017.11.078. Epub 2017 Dec 1. PMID 29452815
- [Derived] Spieth PM, Guldner A, Uhlig C, Bluth T, Kiss T, Schultz MJ, Pelosi P, Koch T, Gama de Abreu M. Variable versus conventional lung protective mechanical ventilation during open abdominal surgery: study protocol for a randomized controlled trial. Trials. 2014 May 2;15:155. doi: 10.1186/1745-6215-15-155. PMID 24885921
- See also: Homepage of the Pulmonary Engineering Group Dresden — http://www.peg-dresden.de